CLINICAL TRIAL: NCT02933151
Title: Health Effects of oraL Protein Supplements in HD (The HELPS-HD Trial) An Open-Label Cluster Randomized Pragmatic Trial Evaluating the Effectiveness of Oral Intradialytic Nutritional Supplements on Mortality in Hemodialysis Patients
Brief Title: Health Effects of oraL Protein Supplements in HD (The HELPS-HD Trial)
Acronym: HELPS-HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dialysis Clinic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HELPS-HD
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Protocol (Other): Facility randomized to follow the usual care nutritional supplement protocol
  Interventions: Dietary Supplement: Nutritional Supplement
- Intensive Protocol (Other): Facility randomized to follow the intensive nutritional supplement protocol
  Interventions: Dietary Supplement: Nutritional Supplement

INTERVENTIONS:
Dietary Supplement: Nutritional Supplement — Selection of which supplement to give to the patients will be left to the dialysis unit's governing body as this study is not interested in a specific supplement's effect on nutrient restoration and subsequent outcomes but rather on oral replacement of amino acids regardless of the agent used.

SUMMARY:
To conduct a pragmatic randomized clinical trial in which the researchers will determine the mortality impact of a protocol whereby all hemodialysis patients receive an oral, protein-based nutritional supplement during the dialysis procedure as compared to the existing nutritional protocol whereby only hemodialysis patients with serum albumin below 3.5 g/dL and incident hemodialysis patients during the first months of care receive an oral, intradialytic protein-based nutritional supplement during the dialysis procedure.

DETAILED DESCRIPTION:
HELPS-HD is a pragmatic, cluster randomized clinical trial comparing the effectiveness of two different oral nutritional supplement protocols and accompanying education. All participants in participating facilities will be asked to participate in the study unless they do not qualify. Reflecting the pragmatic study design targeting broad generalizability, inclusion criteria are broad and exclusions are minimal.

The trial compares Usual Care versus an Intensive Nutritional Supplement Protocol. Facilities are cluster randomized into one of two protocols:

1. Usual care protocol which will continue the current nutritional supplement protocol for all patients at the dialysis facility, whereby those with albumin below 3.5 g/dL receive supplement
2. Intensive nutritional supplement protocol, which will prescribe nutritional supplements for all patients at the dialysis facility regardless of serum albumin levels

The majority of DCI facilities currently have the majority of their patients prescribed the usual care oral nutritional supplement protocol, with 20-30% of patients at any given time receiving an in-center oral nutritional supplement based on either incident hemodialysis status or low serum albumin. Of note, all patients are offered the protocol, but approximately 10-20% refuse the protein supplement, often due to taste and individual preference. Being prescribed the protocol does not affect a patient's ability to consume food or other supplements of their choosing before, during (depending on facility and state regulations) or after dialysis; it simply means that they receive an oral nutritional supplement for consumption during dialysis from the dialysis facility included as a part of their routine dialysis care. The specific nutritional supplement is not specified in the protocol, although many facilities currently use Prostat due to pricing and availability. The protocol prescribes approximately 15 g of oral protein supplement; when Prostat is used, this is accomplished by drinking 30 mL of Prostat. In cases of facility or patient preference, including taste fatigue, other supplements can be used in the current usual care protocol in lieu of Prostat. For example, the PI's facility currently has some patients receiving Prostat while others receive BodyQuest Protein Ice Cream, reflecting patient preference. Nutritional supplements utilized during the trial will vary, but should contain approximately 15 g (range 12 to 20 g) of protein with low sodium, potassium and phosphorus content. Based on current use within DCI and availability as well as prior experiences and cost, the following supplements are anticipated:

1. BodyQuest Protein Ice Cream, which contains 16 g of protein and 120 kcal per serving
2. Prostat, Sugar Free, which contains 15 g of protein and 100 kcal per serving
3. LiquaCel Liquid Protein, which contains 16 g of protein and 90 kcal per serving
4. ZonePerfect Nutrition Bars ( flavor varied to avoid taste fatigue), which contain ~ 15 g of protein and ~ 210 kcal per serving
5. Nepro, which contains 19 g of protein and 425 kcal per serving.

As occurs currently in practice, the serum albumin level from routinely drawn monthly labs will automatically feed into the electronic centralized nutritional supplement prescribing protocols, from which supplements are then prescribed and administered. The DCI electronic oral nutritional supplement protocol will be used in the same manner as in current practice and follow the same rules for dosing and stoppage for the usual care arm, while protocol-based administration will continue regardless of serum albumin level for the intensive protocol arm. All new patients at the time of dialysis initiation (first dialysis session) will receive an oral nutritional supplement if prescribed the protocol by their physician, regardless of intensive or usual care protocol assignment based on their facility. The specific supplement is typically based upon what the individual facility has available and on storage space within facilities. For example, one supplement is a frozen protein supplement (BodyQuest Protein Ice Cream) that can only be used in facilities that have adequate space for food freezers.

As a non-blinded study, the treating physicians will be aware of the study allocation of the facility. In facilities assigned to the intensive oral nutritional supplement intervention, an order will be generated in the DCI MIS by DCI Information Services for administration of an oral protein supplement at each dialysis session. Similarly, in patients assigned to the standard oral nutritional supplement intervention, a renewal order of the current supplement protocol will be generated. As with all orders pertaining to in-center hemodialysis care, the order for intensive versus standard nutritional supplement protocol will need to be signed electronically by the physician caring for the patient. If the physician does not sign this order, the patient will not receive nutritional supplements. The physician, regardless of randomization, can elect to discontinue the supplement order at any time.

As is currently done in practice, the dialysis nurse will record in the treatment record that the nutritional supplement has been dispensed and whether and when it was consumed. Supplements should be distributed and consumed within the first 30 minutes of initiation of a dialysis session.

Within all facilities, patients will receive information regarding the nutritional supplement trial. Educational posters will be displayed in public waiting areas, including signs and posters that inform patients that the site is participating in the trial as well as signs and posters that promote the importance of nutrition and adequate protein intake in recipients of hemodialysis. Every dialysis facility, as a condition for coverage by CMS, is required to have a dietician who provides nutritional information to patients. Regardless of randomization assignment, this individual will continue to encourage appropriate protein intake for dialysis patients, including recommendations for protein and other hemodialysis-appropriate diet consumption at home.

Facilities randomized to usual care and to intensive supplements will have slightly different approaches. First, facilities randomized to the usual care arm will have different signs and posters than those randomized to the intensive arm. Usual care arm materials will promote the need for nutrition and encourage supplement consumption when the albumin is low. Patients are informed of their serum albumin levels monthly at dialysis when they receive feedback from the dietician. In these conversations, the dietician will continue to emphasize protein consumption as per prior routine. For intensive facilities, materials will focus on the catabolic stresses induced by dialysis regardless of baseline albumin level, and emphasize that oral nutritional supplements taken early during dialysis may be able to impact catabolism. Reflecting the open nature of dialysis facilities, if neighboring patients are on different treatment regimens, they are likely to overhear the specific counseling given to other patients and are likely to appreciate that others are receiving more or less supplements than they are. Finally, there is a group mentality prevalent among dialysis patients such that they expect to receive similar treatment and interventions. These factors reinforce the hemodialysis environment as best suited to cluster randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Receipt of in-center hemodialysis in a facility participating in the trial
2. Able to consume oral nutritional supplements
3. Age ≥18 years

Exclusion Criteria:

1. Tube feed or intravenous feed dependent
2. Unable to feed oneself or request help with feeding if a supplement is provided
3. Known allergy to ingredient(s) of the supplement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10457 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Weiner, MD, Principal Investigator — DCI/Tufts
Locations (2):
- United States (2):
  - DCI Jacksonville, Jacksonville, Florida
  - Dialysis Clinic, Inc (Corporate), Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mah JY, Choy SW, Roberts MA, Desai AM, Corken M, Gwini SM, McMahon LP. Oral protein-based supplements versus placebo or no treatment for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2020 May 11;5(5):CD012616. doi: 10.1002/14651858.CD012616.pub2. PMID 32390133

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 10457 patients consented in participating facilities. Because all incident patients, regardless of facility allocation, received an identical nutritional supplement protocol for the first 120 days, incident patients are excluded from analyses for the 1st 120 days. This results in an analytic dataset of 9896 individuals that serves as the basis for Table 1 and all primary analyses.
Units Other Than Participants: Hemodialysis Facilities
Period: Overall Study
Arm/Group | Usual Care Protocol | Intensive Protocol
Started | 4763; 52 Hemodialysis Facilities | 5133; 53 Hemodialysis Facilities
Completed | 2215; 52 Hemodialysis Facilities (No new patients were allocated to the study after December 31, 2019. Intervention was planned through June 30, 2020 for both study groups. Nutritional supplement administration in all DCI clinics ceased on April 8, 2020 due to COVID and a ban on eating in dialysis facilities following mask mandates. This was formally transmitted to all study sites on April 13, 2020. Follow-up for vital status continued through August 2020. Censoring reasons are described below as outcomes are 'completion'.) | 2320; 53 Hemodialysis Facilities (No new patients were allocated to the study after December 31, 2019. Intervention was planned through June 30, 2020 for both study groups. Nutritional supplement administration in all DCI clinics ceased on April 8, 2020 due to COVID and a ban on eating in dialysis facilities following mask mandates. This was formally transmitted to all study sites on April 13, 2020. Follow-up for vital status continued through August 2020. Censoring reasons are described below as outcomes are 'completion'.)
Not Completed | 2548; 0 Hemodialysis Facilities | 2813; 0 Hemodialysis Facilities
Not completed — Lost to Follow-up | 19 | 18
Not completed — Death | 1732 | 1827
Not completed — Transplant | 210 | 278
Not completed — Withdrawal from HD (Death equivalent analytically) | 24 | 29
Not completed — Transferred to PD or a non-DCI facility | 516 | 632
Not completed — Recovered Kidney Function | 47 | 29

BASELINE CHARACTERISTICS:
Population: Primary analyses incorporate a 120 day lag for incident dialysis patients as the usual care and intensive protocols were identical during the time of hemodialysis initiation, such that 9896 participants were in the analytic dataset (4763 in usual care and 5133 in intensive nutritional supplement protocols) received the intervention of a total of 10457 participants allocated to a trial intervention. There were 561 incident hemodialysis patients who did not remain in the DCI facility past day 120.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care Protocol | Intensive Protocol | Total
Number analyzed (Participants) | 4763 | 5133 | 9896
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2357 | 2591 | 4948
  >=65 years | 2406 | 2542 | 4948
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (14.2) | 62.6 (14.8) | 63.0 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2081 | 2248 | 4329
  Male | 2682 | 2885 | 5567
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 183 | 379 | 562
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1648 | 1930 | 3578
  White | 2631 | 2365 | 4996
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 301 | 459 | 760

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: All-cause mortality, assessed from day 0 of study initiation in prevalent patients and day 120 of study initiation in incident patients as all incident patients are provided nutritional supplements during their first 120 days of hemodialysis. Withdrawal from dialysis was classified as death.
  Note that AEs and SAEs were not specifically classified given the minimal risk intervention (protocol prescribing a food containing ~15 g of protein in some participants in usual care facilities and all participants in intensive protocol facilities) and the pragmatic trial design.
Time Frame: Intervention discontinued on April 13, 2020 due to Covid-related prohibition on eating in facilities. Event follow-up concluded on August 13, 2020. Follow-up time varied among participants, with the maximum of approximately 3.5 years.
Population: Incident and prevalent hemodialysis patients at 105 participating hemodialysis facilities in the analytic dataset
Measure: Number; unit: participants
Units Other Than Participants: Hemodialysis Facilities
Arm/Group | Usual Care Protocol | Intensive Protocol
Number analyzed (Participants) | 4763 | 5133
Number analyzed (Hemodialysis Facilities) | 52 | 53
participants | 1756 | 1856
Statistical Analysis 1: Comparison: Usual Care Protocol vs Intensive Protocol; Test type: Superiority; Cox Proportional Hazard = 1.03, 95% CI 2-sided [0.92 to 1.14] — Reference group is usual care

2. Secondary Outcome: Hospitalization
Description: Time to First Hospitalization
Time Frame: Median 7.1 months (25th to 75th percentile: 3.0, 10.9 months)
Population: First hospitalization in the lagged analyses
Measure: Number; unit: Patient level hospitalizations
Units Other Than Participants: Hemodialysis Facilities
Arm/Group | Usual Care Protocol | Intensive Protocol
Number analyzed (Participants) | 4763 | 5133
Number analyzed (Hemodialysis Facilities) | 52 | 53
Patient level hospitalizations | 3655 | 3916

ADVERSE EVENTS:
Time Frame: Median follow-up time was 21.4 months, with a 25th percentile of 10.4 months and a 75th percentile of 37.4 months.
Description: Systematic assessment of mortality and hospitalization. Other events not collected given minimal risk intervention and pragmatic trial design.
  Over the time frame, usual care had 3655 first hospitalizations and the intervention had 3916 first hospitalizations.
Arm/Group | Usual Care Protocol | Intensive Protocol
All-Cause Mortality (participants affected / at risk) | 1732/4763 | 1827/5133
Serious Adverse Events (participants affected / at risk) | 0/4763 | 0/5133
Other Adverse Events (participants affected / at risk) | 0/4763 | 0/5133

LIMITATIONS AND CAVEATS:
Cluster-randomized pragmatic clinical trial with baseline clinical data and outcome ascertainment dependent on clinical data entered into the EHR with resultant less rigorous data capture of adverse events than in non-pragmatic trials and therefore a focus on the all-cause mortality outcome. With the COVID pandemic, nutritional supplements were banned during dialysis in all dialysis facilities in April 2020, resulting in cessation of the trial intervention 3 months earlier than planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT02933151/Prot_SAP_000.pdf